CLINICAL TRIAL: NCT02972710
Title: A Comparison of Two Thoracic Manipulation Techniques to Improve Neck Pain: A Randomized Control Trial
Brief Title: A Comparison of Two Thoracic Manipulation Techniques to Improve Neck Pain
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Arizona University (Other)
Responsible Party: Principal Investigator, Tarang Jain, Assistant Professor - Physical Therapy and Athletic Training, Northern Arizona University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 962801-1
Record Dates: First submitted 2016-11-17; First posted 2016-11-23 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supine thoracic spine manipulation (Active Comparator): Supine thoracic spine thrust manipulation (lying face-up on the treatment table) will be given 2 times at 3 treatment sessions (Weeks 0, 1, and 2)
  Interventions: Other: Supine thoracic spine thrust manipulation
- Seated thoracic spine manipulation (Active Comparator): Seated thoracic spine thrust manipulation will be given 2 times at 3 treatment sessions (Weeks 0, 1, and 2).
  Interventions: Other: Seated thoracic spine thrust manipulation

INTERVENTIONS:
Other: Supine thoracic spine thrust manipulation — The participant will be positioned so that small amplitude quick stretch can be applied to the least mobile area of the thoracic spine that is identified during the spinal segmental mobility testing. The thoracic spine thrust manipulation will be applied at an appropriate range of motion as identified by the clinician.
  Arms: Supine thoracic spine manipulation
Other: Seated thoracic spine thrust manipulation — The participant will be positioned so that small amplitude quick stretch can be applied to the least mobile area of the thoracic spine that is identified during the spinal segmental mobility testing. The thoracic spine thrust manipulation will be applied at an appropriate range of motion as identified by the clinician.
  Arms: Seated thoracic spine manipulation

SUMMARY:
The purpose of this study is to compare the short-term effects of two different thoracic spine thrust manipulation techniques on neck range-of-motion, pain, and self-reported disability in individuals experiencing neck pain.

DETAILED DESCRIPTION:
The study will be conducted at the Musculoskeletal clinical facility in the Dept. of Physical Therapy and Athletic Training, Northern Arizona University, Flagstaff AZ. The investigators aim to test a maximum of 76 participants in this study. A phone screening will determine initial eligibility. If the participant meets the inclusion criteria and is not excluded after the phone screen, an appointment will be scheduled. Final eligibility will be determined in the initial session after the participant completes the outcome measures and is evaluated by a licensed physical therapist.

Participants will be involved in the study over a 4 week period. Each participant will be asked to attend 4 sessions, with one week in between each session as follows: Week 0 = baseline assessment and treatment 1; Week 1= treatment 2; Week 2 = treatment 3; and week 4 = follow-up assessment.

After completion of the baseline assessment, qualified participants will be randomly assigned to either a supine or prone thoracic spine thrust manipulation intervention.

ELIGIBILITY:
Inclusion Criteria:

* Between 20 and 50 years of age (inclusive)
* Primary complaint of neck pain with or without symptoms that spread down into one arm
* Overall rating of neck pain intensity is at least 3/10; the overall rating is the average of the participant's rating of current, least, and worst pain experienced over the previous 24 hours on separate numeric pain rating scales where 0 corresponds to "no pain" and 10 corresponds to "worst possible pain"
* Neck Disability Index (NDI) score > 10 points (measure of self-reported disability with a 0 to 50-point scale where higher scores indicate higher levels of disability)
* Proficient in speaking and reading English to complete outcome questionnaires

Exclusion Criteria:

* Neck pain related to a motor vehicle accident or other trauma within the previous 6 weeks
* Neck pain that spreads down into both arms
* Low back pain or thoracic origin of pain
* Nerve root involvement; defined as the presence of two or more neurological findings (e.g., decreased strength, diminished deep tendon reflex, or decreased sensation) at the same nerve root level
* Diagnosis of cervical spinal stenosis (narrowing of the central canal that contains the spinal cord)
* History of spinal tumors, spinal infection, cervical spine fracture, or previous neck surgery
* Pending legal action related to current episode of neck pain
* Contraindications to thoracic spine thrust manipulation

  1. serious pathologies or conditions (tumor, fracture, metabolic diseases, rheumatoid arthritis, osteoporosis, history of prolonged steroid use)
  2. hyperreflexia
  3. unsteadiness during gait
  4. nystagmus
  5. loss of visual acuity
  6. impaired sensation of the face
  7. altered taste
  8. the presence of pathological reflexes
  9. pregnancy or considering pregnancy

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale (NPRS) | Change in NPRS scores at different time points (Baseline (Week 0) during initial visit before 1st treatment, Week 1, Week 2, and Week 3)
  Each participant's neck pain intensity will be assessed by use of the Numeric Pain Rating Scale (NPRS of 0-10)
Neck Range of Motion | Change in Neck ROM at different time points (Baseline (Week 0) during initial visit before 1st treatment, Week 1, Week 2, and Week 3)
  Cervical range of motion measured with the Goniometer
Neck Disability Index (NDI) | Change in NDI at different time points (Baseline (Week 0) during initial visit before 1st treatment, Week 1, Week 2, and Week 3)
  The Neck Disability Index (NDI) is a self-reported measure of disability consisting of a 0-50 point scale where higher scores indicate higher levels of disability
Shortened version of the Disabilities of the Arm, Shoulder, and Hand questionnaire (Quick DASH) | Change in QuickDASH scores at different time points (Baseline (Week 0) during initial visit before 1st treatment, Week 1, Week 2, and Week 3)
  The shortened version of the Disabilities of the Arm, Shoulder, and Hand (Quick DASH) questionnaire is a self-report measure of function that can assess how neck pain may be impacting daily activities that require use of the upper limb

CONTACTS AND LOCATIONS:
Overall Officials: John Heick, PT, PhD, DPT, Principal Investigator — Northern Arizona University
Locations (1):
- Northern Arizona University, Flagstaff, Arizona, United States

IPD SHARING:
Plan to Share IPD: No